CLINICAL TRIAL: NCT03326271
Title: Postoperative Periprosthetic Fractures in Hip Fracture Patients: Comparison of the Exeter Stem and the Anatomic SP2 Lubinus Stem
Brief Title: Postoperative Periprosthetic Fractures in Hip Fracture Patients: Exeter vs Anatomic SP2 Lubinus Stem
Acronym: PPFEvL
Status: Completed | Type: Observational
Sponsor: Sundsvall Hospital (Other)
Collaborators: Sunderby Hospital (Other); Karolinska Institutet (Other)
Responsible Party: Sponsor
Other Study IDs: Multicenter_PPF
Record Dates: First submitted 2017-10-11; First posted 2017-10-31 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Femoral Neck Fractures; Periprosthetic Fractures
MeSH Terms: conditions — Femoral Neck Fractures; Periprosthetic Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lubinus SP2 stem: Patients treated with a cemented Lubinus SP2 stem for a femoral neck fracture. Both total hip arthroplasty and hemiarthroplasty are included.
  Interventions: Procedure: Lubinus SP2 stem
- Exeter stem: Patients treated with a cemented Exeter stem for a femoral neck fracture. Both total hip arthroplasty and hemiarthroplasty are included.
  Interventions: Procedure: Exeter stem

INTERVENTIONS:
Procedure: Exeter stem — Patients treated with an total or hemiarthroplasty using a Exeter stem for a displaced femoral neck fracture
  Groups: Exeter stem
Procedure: Lubinus SP2 stem — Patients treated with an total or hemiarthroplasty using a SP2stem for a displaced femoral neck fracture
  Groups: Lubinus SP2 stem

SUMMARY:
Recent studies have indicated a high incidence of postoperative periprosthetic femoral fracture in elderly patients treated with two commonly used cemented polished, tapered femoral stems. The aim of this study was to compare the prevalence and incidence rate of PPF in a cohort of elderly with femoral neck fractures (FNF) treated with either a collarless, polished, tapered stem (Exeter) or an anatomic matte stem (Lubinus SP 2).

Patients and Methods In a multicentre retrospective cohort study 2529 patients 60 years and above, with a FNF as indication for primary surgery with a cemented hip arthroplasty were included. Patients were treated either with a polished tapered Exeter stem or a matte anatomic Lubinus SP12 stem according to the surgeons preference or to the praxis of the present department.

The incidence of perprosthetic femoral fractures Hip-related complications and repeat surgery were assessed at a minimum follow-up of 2 years postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Femoral neck fracture
* Treated with hip arthroplasty with Exeter or SP2 stem

Exclusion Criteria:

* Patological fracture
* Other typ of stem

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients at above mentioned centers presented with a femoral neck fracture treated with hip arthroplasty between 2006-2014 were followed 2017 or until death.
Sampling Method: Non-Probability Sample
Enrollment: 2527 (Actual)
Dates: Start 2016-05-04 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-10-11 (Actual)

PRIMARY OUTCOMES:
Periprosthetic femoral fractures | 2006-2014
  The incidence of postoperative periprosthetic femoral fractures are compared between the two groups studied (patients treated with Exeter stem or Lubinus SP2 stem. The hypothesis that the type of stem affects the incidence of periprosthetic femoral fractures are studied. The comparison will be analysed using cox proportional hazards or poisson regression analysis.

SECONDARY OUTCOMES:
Riskfactors for periprosthetic fractures | 2006-2014
  Sex (male or female), age (years), ASA class (1-2 or 3-4), Exeter stem size (0-2, 3-4, 5-6) and surgical approach (direct lateral or posterolateral) type of stem used (Lubinus Sp2 or Exeter stem)

IPD SHARING:
Plan to Share IPD: No
No individual data are presented.

REFERENCES:
- [Background] Inngul C, Enocson A. Postoperative periprosthetic fractures in patients with an Exeter stem due to a femoral neck fracture: cumulative incidence and surgical outcome. Int Orthop. 2015 Sep;39(9):1683-8. doi: 10.1007/s00264-014-2570-0. Epub 2014 Oct 24. PMID 25341951
- [Background] Mukka S, Mellner C, Knutsson B, Sayed-Noor A, Skoldenberg O. Substantially higher prevalence of postoperative peri-prosthetic fractures in octogenarians with hip fractures operated with a cemented, polished tapered stem rather than an anatomic stem. Acta Orthop. 2016 Jun;87(3):257-61. doi: 10.3109/17453674.2016.1162898. Epub 2016 Apr 4. PMID 27045318
- [Background] Broden C, Mukka S, Muren O, Eisler T, Boden H, Stark A, Skoldenberg O. High risk of early periprosthetic fractures after primary hip arthroplasty in elderly patients using a cemented, tapered, polished stem. Acta Orthop. 2015 Apr;86(2):169-74. doi: 10.3109/17453674.2014.971388. Epub 2014 Oct 3. PMID 25280133
- [Background] Mardian S, Perka C, Schaser KD, Gruner J, Scheel F, Schwabe P. Cardiac disease and advanced age increase the mortality risk following surgery for periprosthetic femoral fractures. Bone Joint J. 2017 Jul;99-B(7):921-926. doi: 10.1302/0301-620X.99B7.BJJ-2016-0974.R1. PMID 28663398
- [Derived] Mellner C, Mohammed J, Larsson M, Esberg S, Szymanski M, Hellstrom N, Chang C, Berg HE, Skoldenberg O, Knutsson B, Morberg P, Mukka S. Increased risk for postoperative periprosthetic fracture in hip fracture patients with the Exeter stem than the anatomic SP2 Lubinus stem. Eur J Trauma Emerg Surg. 2021 Jun;47(3):803-809. doi: 10.1007/s00068-019-01263-6. Epub 2019 Nov 18. PMID 31740996